CLINICAL TRIAL: NCT06374160
Title: Better Symptom Control With Exercise in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Exercise in Patients With Advanced Non-small Cell Lung Cancer
Acronym: BREATH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 70115371
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Advanced Lung Carcinoma; First Line Treatment; Second Line Treatment; NSCLC Stage IV; NSCLC Stage IIIB; Palliative Treatment; NSCLC Stage IIIC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: BREATH is a prospective 3-arm 2:1:1 randomized controlled trial (RCT). The first arm represents the control group, which will receive the standard treatment for the first 12 weeks (recommendations for physical activity during cancer treatment). The other two arms represent the exercise groups, one group will receive individualized endurance training and the other group a combination of individualized endurance and strength training. All arms will be treated for 12 weeks. Afterwards, the patients in the control group are randomized to one of the other two study arms and then also treated twice for 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (endurance training + strength training) (Experimental): Frequency: 2 supervised exercise sessions per week.
  Session Breakdown:
  Duration: 60 minutes per session. Aerobic Endurance Training: 20 minutes. Strength Training: 40 minutes.
  Aerobic Interval Training:
  Set at 50% of maximal workload based on spiroergometry. Five sets of 2 minutes of exertion; 5 sets of 1 minute of recovery; Total exertion time: 20 minutes
  Strength Training:
  Muscle Groups Targeted: Major muscle groups. Sets and Repetitions: 2 sets with 8-12 repetitions.
  Training Intensity:
  Range: 50-80% of 1-RM (1-repetition maximum)
  Interventions: Behavioral: Exercise intervention
- Arm B (endurance exercise) (Experimental): Frequency: 2 supervised exercise sessions per week.
  Session Breakdown:
  Duration: Approximately 30 minutes. Focus: Aerobic endurance training. Followed by 10 minutes of Respiratory therapy.
  Endurance Training:
  Method: Intervals for a balance between exertion and recovery. Intensity: Set at 50% of maximal workload based on spiroergometry.
  Interventions: Behavioral: Exercise intervention
- Arm C (Usual Care) (No Intervention): The control group receives a one-time sports consultation with general information about daily activities and sports participation, as well as individual training recommendations. After the 12 weeks, the control group will be randomized into one of the exercise therapies.

INTERVENTIONS:
Behavioral: Exercise intervention — Exercise
  Arms: Arm A (endurance training + strength training); Arm B (endurance exercise)

SUMMARY:
Lung cancer is one of the most common types of cancer in Germany, with 56,839 new cases and 45,072 deaths annually. Approximately 70% of patients with non-small cell lung cancer (NSCLC) are diagnosed at an advanced stage and suffer from comorbidities and symptoms such as fatigue, tiredness, and loss of strength. The standard first-line treatment for metastatic NSCLC includes platinum-based chemoimmunotherapy followed by immunotherapy maintenance. Exercise can have positive effects on symptoms such as shortness of breath, fatigue, quality of life, and physical fitness. However, there is a lack of current scientific evidence for the effectiveness of exercise in advanced lung cancer patients. No current trial investigated exercise in advanced NSCLC receiving immunotherapy so far.

The BREATH-study is a prospective 3-arm randomized controlled trial (RCT). In total, the investigators plan to recruit 104 patients. A 2:1:1 randomization will be performed with three study groups: a control group and two exercise therapy groups (strength+endurance exercise/only endurance exercise). One group receives individual endurance training and the other group a combination of individual endurance and strength training. Both treatment groups will be treated twice a week for 12 weeks. The control group will initially receive standard treatment without exercise for 12 weeks and will then be randomized into one of the other two study groups with exercise twice a week for 12 weeks. This approach allows for a sufficiently large sample for comparisons between exercise therapy and the control group, as well as between the two exercise therapy approaches.

The primary aim is to investigate the impact of exercise on V02peak. Secondarily endpoints aim to investigate changes in physical function, patient related outcomes and cardiac function before and after exercise.

ELIGIBILITY:
Inclusion Criteria

* Patients with histologically confirmed non-small cell lung carcinoma in UICC stages IIIB and IV
* First- or second-line therapy (inclusion up to 28 days after the first cycle) in palliative intention
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria

* Severe cardiopulmonary disease (EF<30%)
* Newly occurring or progressive uncontrolled CNS (central nervous system) metastases
* Expected life expectancy < 3 months
* Bone metastases with acute risk of fracture
* ECOG (Eastern Cooperative Oncology Group) performance status > 2
* Acute pulmonary embolism
* Acute myocardial infarction
* Requiring surgery for aortic aneurysm
* Tension pneumothorax
* Lack of proficiency in the German language
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximum oxygen uptake (VO2 peak [ml/min/kg]) | assessed at Baseline, after 12 weeks and 24 weeks of enrolment
  The primary goal is to achieve an improvement in performance (VO2 peak[ml/min/kg]) from T0 (enrolment) to T1 (12 weeks) through exercise compared to the standard treatment. The one-sided alternative hypothesis of a larger improvement in the two treatment groups compared to the control group will be tested statistically as a confirmatory analysis.

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy - Fatigue (FACT-F) | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  The FACT-F is a 13-item questionnaire to assess fatigue in cancer patients. Subscale are physical well-being, social/family well-being, emotional well-being, functional well-being and the fatigue subscale. Based on the subscale the FACIT-F trial outcome index (TOI) Score range 0-108, FACT-G total score (Score range 0-108) and FACIT-F total score (Score range 0-160) can be calculated. The higher the score, the better the Quality of Life.
European Organisation for Research and Treatment of Cancer (EORTC QLQ C30) | assessed at baseline after 12 weeks and 24 weeks of enrolment
  The EORTC QLQ Core Questionnaire is a 30-item instrument meant to assess some of the different aspects that define the quality of life of cancer patients (e.g., physical function, emotional function, symptom scales, and Quality of Life). High scores for functional scales (score 0-100) represent a high level of functioning, high scores for the global health status represent a high quality of life (score 0-100), high scores for symptom scales (score 0-100) represent a high level of symptomatology.
European Organisation for Research and Treatment of Cancer Lung cancer module (EORTC-LC13) | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  The LC13 is a modular supplement to the EORTC-C30 for assessment of symptoms in clinical lung. cancer trials. The scoring range is between 0 to 100, a high score indicating a high level of symptomatology.
Arterial blood pressure | assessed at Baseline, after 12 weeks and 24 weeks of enrolment
  Change during study participation (mmHg)
Change in ECG | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  Changes in 12-lead resting ECG, including PQ [ms], QRS [ms], and QT [ms] intervals
Adherence to exercise intervention | Through study completion, an average of 12 weeks
  The exercise physiologist monitored adherence to the supervised sessions. Based on the absolute numbers of scheduled exercise sessions, both absolute and percentage-based adherence can be calculated and compared between study arms.
Drop-out rate | Through study completion, an average of 12 weeks
  All withdrawals will be considered as dropouts, with reasons noted. Compare the total number of dropouts in each study arm. This provides a straightforward comparison of the raw dropout counts between groups. Also, calculate the percentage of participants who dropped out in each study arm relative to the total number of participants initially assigned to that arm. This allows for a comparison of dropout rates relative to the initial sample size and compared between study arms.
Recruitment rate | At Baseline
  The recruitment rate quantifies the speed of participant enrollment for a study.
Serious Adverse Event/Adverse Events | Through study completion, an average of 12 weeks
  Safety analyses will be based on Adverse Events (AEs), Serious Adverse Events (SAEs) after the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Therapy response | Baseline and after 12 weeks
  Therapy response in the next computer tomography (analogous to RECIST v1.1)
Treatment Toxicity | assessed at baseline after 12 weeks and 24 weeks of enrolment
  Treatment toxicity encompasses the adverse effects experienced by individuals undergoing chemotherapy and exercise regimens concurrently. These effects may manifest as physical symptoms such as fatigue, nausea, muscle weakness, and decreased immune function, which can impact overall well-being and treatment adherence. Monitoring and managing toxicity levels are crucial to ensure patient safety and optimize treatment outcomes. Additionally, integrating exercise interventions alongside chemotherapy may pose unique challenges, as physical activity can exacerbate certain side effects or interact with treatment efficacy. Therefore, careful monitoring and personalized exercise prescriptions are essential to mitigate toxicity risks and enhance the overall tolerability and effectiveness of combined therapy approaches. Toxicity will be reported with CTCAE v5.0
Treatment scheme | assessed at baseline after 12 weeks and 24 weeks of enrolment
  Change in dose or frequency during trial participation
NT-pro-BNP | Up to 24 weeks
  Concentration of N-terminal prohormone of brain natriuretic peptide (NT-pro-BNP), measured in picograms per milliliter (pg/mL) of blood
High sensitive troponin I | Up to 24 weeks
  Concentration of troponin I in nanograms per milliliter [ng/mL] of blood.
Erythrocytes | Up to 24 weeks
  The amount of Erythrocytes per liter [/pl]
Hemoglobin | Up to 24 weeks
  Concentration of hemoglobin in the blood, measured in grams per deciliter (g/dL)
Leukocytes | Up to 24 weeks
  Count of leukocytes per nanoliter [ /nl]
Lymphocytes | Up to 24 weeks
  Count of lymphocytes per nanoliter [ /nl]
Neutrophils | Up to 24 weeks
  Count of neutrophils per nanoliter [ /nl]
CRP | Up to 24 weeks
  Concentration of C-reactive protein (CRP) in the blood, measured in milligrams per deciliter [mg/dL]
CYRFRA 21-1 | Up to 24 weeks
  Concentration of cytokeratin-19 fragment (CYFRA 21-1) in nanograms per milliliter [ng/mL] of blood
Physical function (Hypothetical One-repetition maximum) | assessed at baseline after 12 weeks and 24 weeks of enrolment
  Leg press [kg.], Latissimus pulldown [kg.], bench press [kg.], Crunch [kg.], Leg curl [kg.], Back extension [kg.]
Blood gas analysis pH value | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  pH value
Blood gas analysis (PAO2) | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  Partial pressure of oxygen in arterial blood (PAO2 [mmHg])
Blood gas analysis (SaO2) | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  Arterial oxygen saturation, measured as a percentage (SaO2 [%])
Blood gas analysis (PCO2) | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  Partial pressure of carbon dioxide in arterial blood PCO2 [mmHg]
Blood gas analysis (BE) | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  Base excess (BE) represents the amount of excess or deficit of base (primarily bicarbonate, HCO3-) in the blood [mmol/l]
Blood gas analysis (HCO3) | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  Bicarbonate concentration in the blood HCO3 [mmol/l]
Blood gas analysis (SBCe) | assessed at baseline, after 12 weeks and 24 weeks of enrolment
  Bicarbonate Concentration in the extracellular fluid SBCe [mmol/l]

CONTACTS AND LOCATIONS:
Overall Officials: Mitra Tewes, PD. Dr., Principal Investigator — Department of Palliative Medicine, University Hospital Essen
Locations (1):
- West German Cancer Center (Department of Palliative medicine and Department of Medical Oncology), University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
We will publish a study protocol, including the statistical analysis plan, at an international peer-reviewed journal

REFERENCES:
- [Derived] De Lazzari N, Wiesweg M, Gotte M, Franco J, Mincu RI, Jager J, Huessler EM, Kuklik N, Stang A, Totzeck M, Tewes M. Improving aerobic capacity in patients with advanced non-small cell lung cancer: study protocol of the 3-armed randomized controlled BREATH trial. Trials. 2026 Jan 17. doi: 10.1186/s13063-025-09416-2. Online ahead of print. PMID 41546104